CLINICAL TRIAL: NCT06005675
Title: User Acceptability Evaluation of Pseudophakic Patients Previously Implanted With the TECNIS Odyssey IOL
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIOL111MOLS
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intervention — No study treatments will be administered during this study.

SUMMARY:
Prospective collection of data from medical records, multicenter, post-market clinical follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Previously bilaterally implanted with TECNIS Odyssey IOL, following cataract extraction;
2. Enrollment at least 21 days after second eye surgery;
3. Clear intraocular media in each eye;
4. Signed informed consent and data protection documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries;
5. Availability, willingness, ability, and sufficient cognitive awareness to comply with examination procedures;
6. Ability to understand, read, and write in English

Exclusion Criteria:

1. Concurrent participation in an interventional clinical trial during the time from which the data will be collected;
2. Use of systemic or ocular medication that may affect vision
3. Prior corneal refractive surgery in each eye (i.e., LASIK, PRK, SMILE, RK, CK); NOTE: Limbal relaxing incisions (LRI) are permissible as planned at the time of surgery (intraoperatively) but not postoperatively until after completion of the study visits;
4. Ongoing adverse events that might impact study measurements, as determined by the investigator;
5. Acute or chronic disease or condition, ocular trauma, or surgery that may confound study measurements (e.g., clinically significant macular degeneration, glaucoma, cystoid macular edema, proliferative diabetic retinopathy, keratoconus, etc.);
6. Amblyopia, strabismus, nystagmus in each eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bilateral pseudophakic subjects previously implanted with the TECNIS Odyssey IOL
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Acuities | 1-month postoperative
  Visual Acuity will be collected via observed case data in units of logMAR.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson, Surgical Vision Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (4):
- United States (4):
  - Empire Eye and Laser Center, Bakersfield, California
  - Center For Sight, Venice, Florida
  - Waring Vision Institute, Mt. Pleasant, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu